CLINICAL TRIAL: NCT02187471
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study of DS-5565 for Treatment of Pain Associated With Fibromyalgia
Brief Title: Treatment of Pain Associated With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS5565-A-E310; 2013-005162-20 (EudraCT Number)
Record Dates: First submitted 2014-07-08; First posted 2014-07-11 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pain Associated With Fibromyalgia
Keywords: pain; fibromyalgia
MeSH Terms: conditions — Pain; Fibromyalgia | interventions — mirogabalin; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Participants take one each of placebo tablet and capsule, twice daily (BID)
  Interventions: Drug: Placebo tablet; Drug: Placebo capsule
- Pregabalin (Other): Participants take one pregabalin capsule and one placebo tablet BID
  Interventions: Drug: Pregabalin; Drug: Placebo tablet
- DS-5565 15 mg QD (Experimental): Participants take one each of placebo tablet and capsule in the morning and one placebo capsule in the evening with one DS-5565 tablet once daily (QD)
  Interventions: Drug: DS-5565; Drug: Placebo tablet; Drug: Placebo capsule
- DS-5565 15 mg BID (Experimental): Participants take one placebo capsule with one DS-5565 tablet BID
  Interventions: Drug: DS-5565; Drug: Placebo capsule

INTERVENTIONS:
Drug: DS-5565 — DS-5565 15 mg QD or BID; tablet for oral use
  Other Names: Mirogabalin
  Arms: DS-5565 15 mg BID; DS-5565 15 mg QD
Drug: Pregabalin — Pregabalin capsule for oral use; 75 mg capsule for one week, then 150 mg capsule
  Other Names: Other treatment - not comparator
  Arms: Pregabalin
Drug: Placebo tablet — Placebo tablet for oral use, matching DS-5565 tablet
  Other Names: Tablet Control
  Arms: DS-5565 15 mg QD; Placebo; Pregabalin
Drug: Placebo capsule — Placebo capsule for oral use, matching pregabalin capsule
  Other Names: Capsule Control
  Arms: DS-5565 15 mg BID; DS-5565 15 mg QD; Placebo

SUMMARY:
The main objective of this trial is to compare change in weekly average daily pain score (ADPS) from baseline to Week 13 in participants receiving either dose of DS-5565 versus placebo.

Weekly ADPS is based on daily pain scores reported by the subject that best describes his or her worst pain over the previous 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to give written informed consent
* Able to complete subject-reported questionnaires per the investigator's judgment
* At screening, subjects must meet the 1990 American College of Rheumatology (ACR) criteria for FM, i.e. widespread pain present for at least 3 months and pain in at least 11 of 18 specific tender point sites. In addition, the 2010 ACR criteria must be met:
* Widespread pain index (WPI) ≥ 7 and symptom severity (SS) scale score ≥ 5, or WPI 3 to 6 and SS scale score ≥ 9
* Symptoms have been present at a similar level for at least 3 months
* The subject does not have a disorder that would otherwise explain the pain
* ADPS of ≥ 4 on the 11-point numeric rating scale (NRS) over the past 7 days prior to randomization (based on completion of at least 4 daily pain diaries during the 7-day baseline period prior to randomization)
* Subject must have documented evidence of a fundoscopic examination (with pupil dilation) within 12 months prior to screening or at screening.
* Women of child-bearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy during the study and for 4 weeks after study completion.

Exclusion Criteria:

* Clinically significant unstable neurologic, psychiatric, ophthalmologic, hepatobiliary, respiratory, or hematologic illness or unstable cardiovascular disease (e.g. severe hypotension, uncontrolled cardiac arrhythmia, or myocardial infarction) or any other concurrent disease within 12 months prior to screening that in the opinion of the investigator would interfere with study participation or assessment of safety and tolerability
* Anticipation of initiation or significant change to normal daily exercise routines or need for ongoing use of concomitant medications or non-pharmacological pain management techniques that may confound assessments of efficacy and/or safety
* Unable to undergo pre-study washout of prohibited concomitant medications
* Subjects who are at risk of suicide as defined by their responses to the Columbia-Suicide Severity Rating Scale (C-SSRS) or in the opinion of the investigator. Note: Patients answering "yes" to any of the C-SSRS questions at screening must be excluded. Such patients should be referred immediately to a mental health professional for appropriate evaluation.
* Current severe or uncontrolled major depressive disorder or anxiety disorders as assessed by the Mini-international Neuropsychiatric Interview (MINI) mild to moderate major depression or anxiety disorders are permitted provided that the investigator assesses the patient as clinically stable and appropriate for entry into the study.
* Any diagnosis of lifetime bipolar disorder or psychotic disorder
* Subjects with pain due to other conditions (e.g. diabetic peripheral neuropathic pain or post-herpetic neuralgia) that in the opinion of the investigator, would confound assessment or self-evaluation of the pain associated with FM.
* Subjects with pain due to any widespread inflammatory musculoskeletal disorder (e.g. rheumatoid arthritis, lupus) or widespread rheumatic disease other than FM.
* Abuse or dependence of prescription medications, street drugs, or alcohol within the last 1 year
* Any history of a malignancy other than basal cell carcinoma within the past 5 years
* A diagnosis of untreated sleep apnea or initiation of treatment for sleep apnea within the past 3 months
* Pregnancy or breast-feeding, or intent to become pregnant during the study period
* Subject is currently enrolled in or has not yet completed at least 30 days since ending another investigational device or drug study or is receiving other investigational agents.
* Known hypersensitivity to alpha2-delta (α2δ) ligands or other components of the study medications. Note: Prior exposure to DS-5565 is allowed, as long as hypersensitivity to DS-5565 was not observed.
* Subjects who are unlikely to comply with the protocol (e.g. uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the investigator to be unlikely to complete the study.
* Abnormal investigative tests (i.e. electrocardiograms [ECGs]) and laboratory values judged by the investigator to be clinically significant at screening, with particular focus on: a. Abnormal renal function defined as calculated creatinine clearance (CrCl) < 60 mL/min determined by the central laboratory using the modified Cockcroft-Gault equation; blood urea nitrogen> 1.5 × upper limit of normal (ULN); creatine kinase > 3.0 × ULN; serum creatinine > 1.6 mg/dL (> 141.4 μmol/L); b. Abnormal liver function defined as aspartate aminotransferase (AST) > 2.0 × ULN, alanine aminotransferase (ALT) > 2.0 × ULN; alkaline phosphatase > 1.5 × ULN; total bilirubin> 1.2 × ULN. If a subject has total bilirubin > 1.2 ULN, unconjugated and conjugated bilirubin fractions should be analyzed and only subjects documented to have Gilbert's syndrome may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1301 (Actual)
Dates: Start 2015-01-16 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (153):
- United States (90):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Covina, California
  - El Cajon, California
  - Encino, California
  - Huntington Beach, California
  - Lakewood, California
  - Lomita, California
  - Los Angeles, California
  - National City, California
  - Northridge, California
  - Oceanside, California
  - Sacramento, California
  - Upland, California
  - Walnut Creek, California
  - Boca Raton, Florida
  - DeLand, Florida
  - Edgewater, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Largo, Florida
  - Lauderdale Lakes, Florida
  - Maitland, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sunrise, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Winter Haven, Florida
  - Winter Park, Florida
  - Dawsonville, Georgia
  - Marietta, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Evansville, Indiana
  - Granger, Indiana
  - Overland Park, Kansas
  - Owensboro, Kentucky
  - Lake Charles, Louisiana
  - New Orleans, Louisiana
  - Frederick, Maryland
  - Brockton, Massachusetts
  - North Dartmouth, Massachusetts
  - Ann Arbor, Michigan
  - Lansing, Michigan
  - Rochester Hills, Michigan
  - Florissant, Missouri
  - Hazelwood, Missouri
  - O'Fallon, Missouri
  - Bellevue, Nebraska
  - Newington, New Hampshire
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Cedarhurst, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Minot, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Media, Pennsylvania
  - Wyomissing, Pennsylvania
  - Greenville, South Carolina
  - Mt. Pleasant, South Carolina
  - Chattanooga, Tennessee
  - Franklin, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Richland, Washington
- Argentina (10):
  - CABA, Buenos Aires
  - La Plata, Buenos Aires
  - Lanús, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Quilmes, Buenos Aires
  - San Fernando, Buenos Aires
  - Rosario, Santa Fe Province
  - Córdoba
  - San Miguel de Tucumán
  - Santa Fe
- Austria (3):
  - Klagenfurt
  - Senftenberg
  - Vienna
- Belarus (2):
  - Minsk
  - Vitebsk
- Belgium (4):
  - Brussels
  - Edegem
  - Gozée
  - Oostham
- Chile (4):
  - Antofagasta
  - Providencia
  - Puerto Varas
  - Viña del Mar
- Colombia (2):
  - Barranquilla
  - Bogotá
- Israel (4):
  - Haifa
  - Kfar Saba
  - Ramat Gan
  - Tel Aviv
- Mexico (5):
  - Cuautitlán Izcalli
  - Durango
  - Guadalajara
  - León
  - Mexico City
- Poland (10):
  - Elblag
  - Gdansk
  - Katowice
  - Krakow
  - Lublin
  - Nadarzyn
  - Nowa Sól
  - Torun
  - Tychy
  - Warsaw
- Portugal (7):
  - Aveiro
  - Braga
  - Guimarães
  - Lisbon
  - Ponte de Lima
  - Porto
  - Vila Nova de Gaia
- Slovenia (2):
  - Ljubljana
  - Slovenj Gradec
- Spain (8):
  - Alicante
  - Barcelona
  - Elche
  - Granada
  - Guadalajara
  - Madrid
  - Santiago de Compostela
  - Seville
- Switzerland (2):
  - Geneva
  - Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Arnold LM, Whitaker S, Hsu C, Jacobs D, Merante D. Efficacy and safety of mirogabalin for the treatment of fibromyalgia: results from three 13-week randomized, double-blind, placebo- and active-controlled, parallel-group studies and a 52-week open-label extension study. Curr Med Res Opin. 2019 Oct;35(10):1825-1835. doi: 10.1080/03007995.2019.1629757. Epub 2019 Jul 9. PMID 31284771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2526 participants who met all inclusion criteria and no exclusion criteria were enrolled from 16 Jan 2015 to 12 Jan 2017 at 182 sites. Of the 2526 participants enrolled, 1301 were randomized to treatment.
Pre-assignment Details: Eligible participants were randomized 1:1:1:1 to either DS-5565 15 mg every day (QD) given orally, DS-5565 15 mg twice daily (BID) given orally, placebo given orally as pregabalin placebo and DS-5565 placebo BID, or pregabalin 150 mg BID.
Groups:
- Placebo: Participants who received oral DS-5565 placebo and pregabalin placebo in the morning and evening.
- Pregabalin 150 mg BID: Participants who received oral DS-5565 placebo and pregabalin 150 mg BID in the morning and evening.
- DS-5565 15 mg QD: Participants who received oral DS-5565 placebo and pregabalin placebo in the morning and DS-5565 15 mg and pregabalin placebo in the evening.
- DS-5565 15 mg BID: Participants who received oral DS-5565 15 mg and pregabalin placebo in the morning and evening.
Period: Overall Study
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Started | 325 | 324 | 326 | 326
Completed | 249 | 242 | 240 | 246
Not Completed | 76 | 82 | 86 | 80
Not completed — Protocol Violation | 4 | 5 | 4 | 4
Not completed — Missing | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 18 | 9 | 13 | 11
Not completed — Adverse Event | 24 | 34 | 44 | 36
Not completed — Withdrawal by Subject | 23 | 29 | 22 | 24
Not completed — Other | 7 | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID | Total
Number analyzed (Participants) | 325 | 324 | 326 | 326 | 1301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 296 | 294 | 294 | 290 | 1174
  >=65 years | 29 | 30 | 32 | 36 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.16) | 49.9 (12.02) | 50.1 (11.22) | 49.0 (12.03) | 49.5 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303 | 302 | 302 | 296 | 1203
  Male | 22 | 22 | 24 | 30 | 98
Region of Enrollment [Number; unit: participants]
  Colombia | 0 | 0 | 1 | 0 | 1
  Argentina | 25 | 25 | 19 | 19 | 88
  United States | 190 | 190 | 190 | 190 | 760
  Belarus | 5 | 2 | 2 | 3 | 12
  Portugal | 8 | 8 | 1 | 5 | 22
  Switzerland | 0 | 0 | 1 | 0 | 1
  Spain | 25 | 25 | 27 | 24 | 101
  Austria | 4 | 4 | 10 | 11 | 29
  Belgium | 5 | 5 | 3 | 2 | 15
  Poland | 20 | 21 | 23 | 22 | 86
  Mexico | 9 | 4 | 9 | 7 | 29
  Slovenia | 4 | 2 | 4 | 1 | 11
  Chile | 7 | 11 | 12 | 15 | 45
  Russia | 7 | 7 | 6 | 7 | 27
  Ukraine | 16 | 20 | 18 | 20 | 74

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 13 in Average Daily Pain Score (ADPS) Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: Average daily pain scores (ADPS) reported by the participant that best describes his or her worst pain over the previous 24 hours. A daily pain score has a scale where 0 = no pain to 10 = worst possible pain. Higher scores indicate a worse outcome. For participants with no Week 13 data, the baseline observation was carried forward (BOCF). The mean (multiple imputation estimate) and standard error (multiple imputation) are reported.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 323 | 319 | 324 | 322
units on a scale | -1.90 (0.135) | -2.64 (0.137) | -2.04 (0.138) | -2.30 (0.136)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.4601, Difference of means; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.52 to 0.23], Standard Error of Mean 0.191
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0350, Difference of means; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.77 to -0.03], Standard Error of Mean 0.190
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0001, Difference of means; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.12 to -0.37], Standard Error of Mean 0.191
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0019, Difference of means; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [0.22 to 0.98], Standard Error of Mean 0.193
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0761, Difference of means; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.04 to 0.72], Standard Error of Mean 0.192

2. Secondary Outcome: Number of Participants Who Answered "Much Improved or Better" in Patient Global Impression of Change at Week 13 Receiving DS-5565, Pregabalin, or Placebo
Description: Patient global impression of change (PGIC) on a 7-point categorical scale, where 1 = very much improved and 7 = very much worse. Higher scores indicate worse outcomes. The number of participants with 'much improved or better' status (≤2) is being reported.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 319 | 324 | 323
Participants | 88 | 145 | 127 | 134

3. Secondary Outcome: Change From Baseline to Week 13 in Average Score on the Fibromyalgia Index Questionnaire (FIQ) in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The total FIQ score is composed of 10 items, with a maximum possible score of 100. The first item contains 11 questions related to physical functioning and are rated on a 4-point Likert-type scale, where 0 indicates 'always' and 3 indicates 'never'. The overall impact items are rated on a 0-7 scale for the number of days that the patient felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. The symptoms items are rated on visual analog scales (0-10 cm), with higher numbers indicated greater symptomatology. Final scores range from 0 (no impairment) to 10 (maximum impairment), where higher scores indicate worse outcome.
  For this outcome, the change in total FIQ score from baseline is being reported. Negative values indicate improvement from baseline in impairment.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 322 | 318 | 323 | 320
units on a scale | -15.02 (1.198) | -19.42 (1.222) | -16.61 (1.215) | -20.44 (1.209)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.3407, Difference of means; Mean Difference (Final Values) = -1.59, 95% CI 2-sided [-4.86 to 1.68], Standard Error of Mean 1.670
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0012, Difference of means; Mean Difference (Final Values) = -5.42, 95% CI 2-sided [-8.69 to -2.15], Standard Error of Mean 1.669
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0083, Difference of means; Mean Difference (Final Values) = -4.39, 95% CI 2-sided [-7.66 to -1.13], Standard Error of Mean 1.665
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0946, Difference of means; Mean Difference (Final Values) = 2.80, 95% CI 2-sided [-0.48 to 6.09], Standard Error of Mean 1.677
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.5384, Difference of means; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-4.30 to 2.24], Standard Error of Mean 1.669

4. Secondary Outcome: Number of Participants Classified As Responders at Week 13 Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The ADPS responder rate was defined a priori as the proportion of participants who met the clinically relevant reductions (ie, ≥30% and ≥50%) in ADPS at Week 13 (baseline observation carried forward) compared to Baseline.
Time Frame: Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 319 | 324 | 323
Participants
  30% Responders | 122 | 144 | 121 | 125
  50% Responders | 68 | 95 | 77 | 89

5. Secondary Outcome: Change From Baseline to Week 13 in Multidimensional Fatigue Inventory (MFI-20) General Fatigue Score Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: MFI is a validated 20-item, self-reported instrument designed to measure fatigue in the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. The respondent is asked to mark an 'X' in 1 of 5 boxes arranged linearly where 1 is 'Yes, that is true' and 5 is 'No, that is not true.' Each subscale consists of 4 items, 2 indicative for fatigue and 2 contraindicative. For the indicative questions, a high score indicates a high fatigue level and low scores indicate a low fatigue levels. Conversely, for the contraindicative questions a high score indicates a low fatigue level and a low score indicates a high fatigue level. Overall, respondents are rated on a scale of 0 (no fatigue) to 7 (high fatigue).
  For this outcome, the change from baseline in MFI-20 general fatigue subscale score is being reported. Negative values indicate an improvement in fatigue.
Time Frame: Baseline up to Week 13 postdose
Population: MFI-20 was assessed in the modified intent-to-treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 307 | 299 | 301 | 300
units on a scale | -1.6 (3.55) | -2.6 (4.00) | -2.4 (3.91) | -3.4 (4.54)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0030, ANCOVA; Difference in least squares means = -0.9, 95% CI 2-sided [-1.5 to -0.3], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = -1.7, 95% CI 2-sided [-2.3 to -1.1], Standard Error of Mean 0.30
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0001, ANCOVA; Difference in least squares means = -1.2, 95% CI 2-sided [-1.7 to -0.6], Standard Error of Mean 0.30
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.3562, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.3 to 0.9], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0862, ANCOVA; Difference in least squares means = -0.5, 95% CI 2-sided [-1.1 to 0.1], Standard Error of Mean 0.30

6. Secondary Outcome: Change From Baseline to Week 13 in Hospital Anxiety and Depression Scale (HADS) Measure Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The HADS questionnaire is a reliable, widely-used self-assessment scale to assess symptoms of anxiety and depression. The instrument consists of 7 questions related to anxiety and 7 related to depression, each rated on a 4-point scale (score of 0 to 3). Scores for anxiety and depression are independently summed to compute HADS-Anxiety and HADS-Depression subscale scores, with ranges from 0 to 21, where higher scores indicate greater severity.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed in the modified intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 299 | 324 | 323
units on a scale
  Change from baseline at Week 13: Anxiety: number analyzed (Participants) | 307 | 299 | 301 | 300
  Change from baseline at Week 13: Anxiety | -1.0 (3.58) | -0.9 (3.81) | -1.0 (3.78) | -1.0 (4.10)
  Change from baseline at Week 13: Depression: number analyzed (Participants) | 307 | 299 | 301 | 300
  Change from baseline at Week 13: Depression | -0.8 (3.67) | -1.0 (4.07) | -1.0 (3.80) | -1.2 (3.69)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Anxiety: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.5183, ANCOVA; Difference in least square means = -0.2, 95% CI 2-sided [-0.7 to 0.4], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Anxiety: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.2669, ANCOVA; Difference in least squares mean = -0.3, 95% CI 2-sided [-0.9 to 0.2], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg BID; Anxiety: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.4630, ANCOVA; Difference in least squares means = -0.2, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Anxiety: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.9280, ANCOVA; Difference in least squares means = 0.0, 95% CI 2-sided [-0.5 to 0.6], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Anxiety: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.7089, ANCOVA; Difference in least squares means = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.28
Statistical Analysis 6: Comparison: Placebo vs DS-5565 15 mg QD; Depression: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0669, ANCOVA; Difference in least squares means = -0.5, 95% CI 2-sided [-1.1 to 0], Standard Error of Mean 0.28
Statistical Analysis 7: Comparison: Placebo vs DS-5565 15 mg BID; Depression: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0081, ANCOVA; Difference in least squares means = -0.8, 95% CI 2-sided [-1.3 to -0.2], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg BID; Depression: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0867, ANCOVA; Difference in least squares means = -0.5, 95% CI 2-sided [-1.0 to 0.1], Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Depression: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.9066, ANCOVA; Difference of least squares means = -0.0, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.29
Statistical Analysis 10: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Depression: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.3509, ANCOVA; Difference in least squares means = -0.3, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.29

7. Secondary Outcome: Change From Baseline to Week 13 in Short Form 36 (SF-36) Measure Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The SF-36 is a generic health survey that asks 36 questions to measure functional health and well-being from the patient's point of view. The SF-36 provides scores for 8 health domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) as well as psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores. Each scale is transformed into a 0-100 scale with each question carrying the same weight. The lower the score indicates more disability (ie, worse outcome).
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed in the modified intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 319 | 324 | 323
units on a scale
  Change from baseline to Week 13:Physical Component: number analyzed (Participants) | 307 | 299 | 301 | 300
  Change from baseline to Week 13:Physical Component | 3.78 (7.22) | 6.46 (8.32) | 5.94 (8.06) | 6.22 (8.46)
  Change from baseline to Week 13: Mental Component: number analyzed (Participants) | 307 | 299 | 301 | 300
  Change from baseline to Week 13: Mental Component | 2.23 (9.54) | 1.97 (10.53) | 1.56 (10.19) | 2.71 (9.67)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Physical Component: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0004, ANCOVA; Difference in least squares means = 2.187, 95% CI 2-sided [0.970 to 3.404], Standard Error of Mean 0.6203
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Physical Component: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference of least squares means = 2.483, 95% CI 2-sided [1.265 to 3.701], Standard Error of Mean 0.6209
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg BID; Physical Component: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = 2.621, 95% CI 2-sided [1.401 to 3.840], Standard Error of Mean 0.6215
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Physical Component: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.4877, ANCOVA; Difference in least squares means = -0.434, 95% CI 2-sided [-1.659 to 0.792], Standard Error of Mean 0.6245
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Physical Component: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.8263, ANCOVA; Difference in least squares means = -0.137, 95% CI 2-sided [-1.364 to 1.089], Standard Error of Mean 0.6252
Statistical Analysis 6: Comparison: Placebo vs DS-5565 15 mg QD; Mental Component: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.7567, ANCOVA; Difference in least squares means = 0.228, 95% CI 2-sided [-1.213 to 1.669], Standard Error of Mean 0.7345
Statistical Analysis 7: Comparison: Placebo vs DS-5565 15 mg BID; Mental Component: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0787, ANCOVA; Difference in least squares means = 0.7349, 95% CI 2-sided [-0.149 to 2.735], Standard Error of Mean 0.7349
Statistical Analysis 8: Comparison: Placebo vs Pregabalin 150 mg BID; Mental Component: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.3516, ANCOVA; Difference in least squares means = 0.7358, 95% CI 2-sided [-0.758 to 2.129], Standard Error of Mean 0.7358
Statistical Analysis 9: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Mental Component: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.5344, ANCOVA; Difference in least squares means = -0.458, 95% CI 2-sided [-1.905 to 0.988], Standard Error of Mean 0.7372
Statistical Analysis 10: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Mental Component: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.4107, ANCOVA; Difference in least squares means = 0.607, 95% CI 2-sided [-0.840 to 2.055], Standard Error of Mean 0.7379

8. Secondary Outcome: Change From Baseline to Week 13 in EuroQol Five Dimensions Questionnaire (EQ-5D) Measure Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The EQ-5D is an instrument that shows high construct validity and responsiveness in patients with chronic pain and has been used specifically in fibromyalgia. The EQ-5D includes a descriptive section with 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with a scale that ranges from 0 (no problems) to 5 (extreme problems). These 5 dimensions are combined into an overall health utilities index, and an numeric rating scale (100 mm visual analog scale) that measures perception of overall health, with 0 indicating worst health and 100 representing best imaginable health. A summary index with a maximum total score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum total score of 1 indicates the best health outcome.
  For this outcome, the change from baseline in total EQ-5D score is being reported. Positive values indicate an improvement in health.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed in the modified intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 307 | 299 | 301 | 300
units on a scale | 0.09 (0.19) | 0.1274 (0.20) | 0.10 (0.19) | 0.11 (0.21)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1394, ANCOVA; Difference in least squares means = 0.0203, 95% CI 2-sided [-0.0066 to 0.0471], Standard Error of Mean 0.01369
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1237, ANCOVA; Difference in least squares means = 0.0211, 95% CI 2-sided [-0.0058 to 0.0480], Standard Error of Mean 0.01369
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0049, ANCOVA; Difference in least squares means = 0.0386, 95% CI 2-sided [0.0117 to 0.0655], Standard Error of Mean 0.01371
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1824, ANCOVA; Difference in least squares means = -0.0184, 95% CI 2-sided [-0.0454 to 0.0086], Standard Error of Mean 0.01378
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.2036, ANCOVA; Difference in least squares means = -0.0175, 95% CI 2-sided [-0.0446 to 0.0095], Standard Error of Mean 0.01378

9. Secondary Outcome: Change From Baseline to Week 13 in Average Daily Sleep Interference Score (ADSIS) Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: Pain-associated sleep interference will be assessed using the Average Daily Sleep Interference Score that utilize electronic daily diaries with an 11-point numeric rating scale (NRS) for pain, ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep, unable to sleep). Higher scores indicate worse outcomes.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 319 | 324 | 323
units on a scale | -1.76 (0.116) | -2.71 (0.116) | -2.31 (0.117) | -2.64 (0.116)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0006, Mixed Models Analysis; Difference in least squares means = -0.56, 95% CI 2-sided [-0.87 to -0.24], Standard Error of Mean 0.162
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in least squares means = -0.88, 95% CI 2-sided [-1.20 to -0.57], Standard Error of Mean 0.160
Statistical Analysis 3: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in least squares means = -0.95, 95% CI 2-sided [-1.27 to -0.63], Standard Error of Mean 0.161
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0158, Mixed Models Analysis; Difference in least squares means = 0.39, 95% CI 2-sided [0.07 to 0.71], Standard Error of Mean 0.162
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.6819, Mixed Models Analysis; Difference in least squares means = 0.07, 95% CI 2-sided [-0.25 to 0.38], Standard Error of Mean 0.161

10. Secondary Outcome: Number of Participants Reporting Optimal Sleep at Week 13 on the Medical Outcomes Study (MOS) Sleep Scale Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The MOS Sleep Scale is a 12-item questionnaire from which the following subscales were derived: sleep disturbance (4 items), quantity of sleep/optimal sleep (1 item), snoring (1 item), awakening due to shortness of breath or due to headache (1 item), sleep adequacy (2 items), and somnolence (3 items). In addition, values for sleep disturbances index (9 items), optimal sleep scale (1 item), and sleep quantity scale (1 item) were determined. Most subscales range from 0 to 100, where higher scores indicate more of the concept begin measured (eg., higher sleep disturbance scores indicate greater sleep disturbances).
Time Frame: Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 319 | 324 | 323
Participants | 78 | 107 | 102 | 119

11. Secondary Outcome: Change From Baseline at Week 13 in the Brief Pain Inventory Short Form (BPI-SF) Measure Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The BPI-SF measures pain severity and interference within the past 24 hours. Items are rated on an 11-point NRS from 0 to 10, where 0 indicates does not interfere and 10 indicates completely interferes. Severity score is the average of the responses to the 4 pain intensity items that assess the Worst/Least/Average pain in the last 24 hours and the Pain Right Now. The individual items being reported (using the same scale as noted above) are Severity, General Activity, Mood, Walking Ability, Normal Work, Relations With Other People, Sleep, and Enjoyment of Life. Percentage relief of treatment pain scale ranges from 100% (complete pain relief) to 0% (no pain relief) and higher percentages indicate better outcome. Interference % is the average of responses for General activity, Mood, Walking ability, Normal work, Relations with other people, Sleep, Enjoyment of life where 0% (no interference) to 100% (completely interferes) and negative (ie. lower) percentages indicate better outcomes.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 319 | 324 | 323
units on a scale
  Worst pain: number analyzed (Participants) | 248 | 240 | 239 | 243
  Worst pain | -1.9 (2.26) | -2.7 (2.78) | -2.2 (2.48) | -2.7 (2.52)
  Least pain: number analyzed (Participants) | 248 | 240 | 239 | 243
  Least pain | -1.5 (2.48) | -2.3 (2.58) | -2.0 (2.43) | -2.1 (2.53)
  Average pain: number analyzed (Participants) | 248 | 240 | 239 | 243
  Average pain | -1.5 (2.11) | -2.3 (2.27) | -2.0 (2.28) | -2.3 (2.39)
  Pain right now: number analyzed (Participants) | 248 | 240 | 239 | 243
  Pain right now | -2.1 (2.44) | -2.8 (2.74) | -2.5 (2.50) | -2.9 (2.72)
  Severity score: number analyzed (Participants) | 248 | 240 | 239 | 243
  Severity score | -1.75 (2.05) | -2.55 (2.35) | -2.16 (2.13) | -2.51 (2.26)
  Percentage of relief by treatment of pain: number analyzed (Participants) | 248 | 240 | 239 | 243
  Percentage of relief by treatment of pain | 23.1 (31.93) | 32.6 (35.39) | 31.8 (32.28) | 36.0 (34.68)
  Interference (%): number analyzed (Participants) | 248 | 240 | 239 | 243
  Interference (%) | -16.19 (21.83) | -23.55 (23.60) | -21.66 (22.29) | -25.97 (23.38)
  General activity: number analyzed (Participants) | 248 | 240 | 239 | 243
  General activity | -1.7 (2.60) | -2.5 (2.87) | -2.3 (2.69) | -2.6 (2.82)
  Mood: number analyzed (Participants) | 248 | 240 | 239 | 243
  Mood | -1.6 (2.83) | -2.1 (2.92) | -1.9 (2.95) | -2.4 (2.95)
  Walking ability: number analyzed (Participants) | 248 | 240 | 239 | 243
  Walking ability | -1.4 (2.66) | -1.7 (2.96) | -1.8 (2.73) | -2.1 (2.66)
  Normal work: number analyzed (Participants) | 248 | 240 | 239 | 243
  Normal work | -1.6 (2.52) | -2.3 (2.93) | -2.1 (2.63) | -2.7 (2.73)
  Relations with other people: number analyzed (Participants) | 248 | 240 | 239 | 243
  Relations with other people | -1.3 (2.89) | -1.9 (3.03) | -1.6 (2.95) | -2.0 (2.97)
  Sleep: number analyzed (Participants) | 248 | 240 | 239 | 243
  Sleep | -2.1 (3.13) | -3.6 (3.13) | -3.1 (3.06) | -3.9 (3.08)
  Enjoyment of life: number analyzed (Participants) | 248 | 240 | 239 | 243
  Enjoyment of life | -1.6 (2.94) | -2.4 (3.06) | -2.3 (2.95) | -2.4 (3.27)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Worst pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference of least squares means = -0.8, 95% CI 2-sided [-1.2 to -0.4], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Worst pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.2005, ANCOVA; Difference of least squares means = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Worst pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0010, ANCOVA; Difference in least squares means = -0.6, 95% CI 2-sided [-1.0 to -0.3], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Worst pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0030, ANCOVA; Difference in least squares means = 0.6, 95% CI 2-sided [0.2 to 1.0], Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Worst pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.3351, ANCOVA; Difference in least squares means = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.19
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 150 mg BID; Least pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = -0.8, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs DS-5565 15 mg QD; Least pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0782, ANCOVA; Difference in least squares means = -0.3, 95% CI 2-sided [-0.7 to 0.0], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs DS-5565 15 mg BID; Least pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0068, ANCOVA; Difference in least squares means = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Least pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0169, ANCOVA; Difference in least squares means = 0.4, 95% CI 2-sided [0.1 to 0.8], Standard Error of Mean 0.19
Statistical Analysis 10: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Least pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1481, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.1 to 0.6], Standard Error of Mean 0.19
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 150 mg BID; Average pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = -0.8, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Placebo vs DS-5565 15 mg QD; Average pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0088, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.17
Statistical Analysis 13: Comparison: Placebo vs DS-5565 15 mg BID; Average pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0005, ANCOVA; Difference in least squares means = -0.6, 95% CI 2-sided [-0.9 to -0.3], Standard Error of Mean 0.17
Statistical Analysis 14: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Average pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0627, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.0 to 0.7], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Average pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.3064, ANCOVA; Difference in least squares means = 0.2, 95% CI 2-sided [-0.2 to 0.5], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 150 mg BID; Pain right now: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = -0.8, 95% CI 2-sided [-1.2 to -0.4], Standard Error of Mean 0.20
Statistical Analysis 17: Comparison: Placebo vs DS-5565 15 mg QD; Pain right now: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0868, ANCOVA; Difference in least squares mean = -0.3, 95% CI 2-sided [-0.7 to 0.0], Standard Error of Mean 0.20
Statistical Analysis 18: Comparison: Placebo vs DS-5565 15 mg BID; Pain right now: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0004, ANCOVA; Difference in least squares means = -0.7, 95% CI 2-sided [-1.1 to -0.3], Standard Error of Mean 0.20
Statistical Analysis 19: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Pain right now: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0271, ANCOVA; Difference in least squares means = 0.4, 95% CI 2-sided [0.1 to 0.8], Standard Error of Mean 0.20
Statistical Analysis 20: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Pain right now: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.6838, ANCOVA; Difference in least squares means = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.20
Statistical Analysis 21: Comparison: Placebo vs Pregabalin 150 mg BID; Severity score: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = -0.791, 95% CI 2-sided [-1.129 to -0.454], Standard Error of Mean 0.1720
Statistical Analysis 22: Comparison: Placebo vs DS-5565 15 mg QD; Severity score: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0552, ANCOVA; Difference in least squares means = -0.330, 95% CI 2-sided [-0.667 to 0.007], Standard Error of Mean 0.1718
Statistical Analysis 23: Comparison: Placebo vs DS-5565 15 mg BID; Severity score: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0004, ANCOVA; Difference in least squares means = -0.612, 95% CI 2-sided [-0.950 to -0.275], Standard Error of Mean 0.1718
Statistical Analysis 24: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Severity score: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0077, ANCOVA; Difference in least squares means = 0.462, 95% CI 2-sided [0.122 to 0.801], Standard Error of Mean 0.1729
Statistical Analysis 25: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Severity score: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.3014, ANCOVA; Difference in least squares means = 0.179, 95% CI 2-sided [-0.161 to 0.518], Standard Error of Mean 0.1730
Statistical Analysis 26: Comparison: Placebo vs Pregabalin 150 mg BID; Relief (%) by treatment of pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = 9.6, 95% CI 2-sided [4.9 to 14.3], Standard Error of Mean 2.40
Statistical Analysis 27: Comparison: Placebo vs DS-5565 15 mg QD; Relief (%) by treatment of pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0004, ANCOVA; Difference in least squares means = 8.5, 95% CI 2-sided [3.8 to 13.2], Standard Error of Mean 2.39
Statistical Analysis 28: Comparison: Placebo vs DS-5565 15 mg BID; Relief (%) by treatment of pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = 10.4, 95% CI 2-sided [5.7 to 15.1], Standard Error of Mean 2.39
Statistical Analysis 29: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Relief (%) by treatment of pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.6449, ANCOVA; Difference in least squares means = -1.1, 95% CI 2-sided [-5.8 to 3.6], Standard Error of Mean 2.41
Statistical Analysis 30: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Relief (%) by treatment of pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.7340, ANCOVA; Difference in least square means = 0.8, 95% CI 2-sided [-3.9 to 5.5], Standard Error of Mean 2.41

12. Secondary Outcome: Proportion of Days a Rescue Medication Was Used Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: Proportion of days with rescue medication intake during the double-blind treatment period equals number of days with rescue medication intake/(date of last study drug administration in the double-blind treatment period) - (date of first study drug administration + 1).
Time Frame: Week 1 to Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: proportion of days
Groups:
- Pregabalin: Participants who received oral DS-5565 placebo and pregabalin 150 mg BID in the morning and evening.
Arm/Group | Placebo | Pregabalin | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 324 | 319 | 324 | 323
proportion of days | 0.23 (0.32) | 0.15 (0.25) | 0.21 (0.31) | 0.16 (0.26)
Statistical Analysis 1: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.4816, ANCOVA; Difference in least squares means = -0.016, 95% CI 2-sided [-0.060 to 0.028], Standard Error of Mean 0.0225
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0044, ANCOVA; Difference in least square means = -0.064, 95% CI 2-sided [-.109 to -0.020], Standard Error of Mean 0.0225
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Test type: Superiority; p = 0.0010, ANCOVA; Difference in least squares means = -0.074, 95% CI 2-sided [-0.119 to -0.030], Standard Error of Mean 0.0226
Statistical Analysis 4: Comparison: Pregabalin vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0094, ANCOVA; Difference in least squares means = 0.059, 95% CI 2-sided [0.014 to 0.103], Standard Error of Mean 0.0226
Statistical Analysis 5: Comparison: Pregabalin vs DS-5565 15 mg BID; Test type: Superiority; p = 0.6527, ANCOVA; Difference in least squares means = 0.010, 95% CI 2-sided [-0.034 to 0.055], Standard Error of Mean 0.0226

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 4 weeks after the last dose of study medication, up to 2 years 3 months.
Description: A TEAE was any adverse event that emerged on or after the first dosing of double-blind study medication and during study treatment up to 4 weeks after the last dose of double-blind study medication (having been absent prior to treatment) or worsened relative to the pre-double-blind treatment state.
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
All-Cause Mortality (participants affected / at risk) | 0/324 | 0/319 | 0/324 | 0/323
Serious Adverse Events (participants affected / at risk) | 9/324 | 2/319 | 5/324 | 5/323
Other Adverse Events (participants affected / at risk) | 171/324 | 289/319 | 258/324 | 247/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=324) | Pregabalin 150 mg BID (N=319) | DS-5565 15 mg QD (N=324) | DS-5565 15 mg BID (N=323)
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=324) | Pregabalin 150 mg BID (N=319) | DS-5565 15 mg QD (N=324) | DS-5565 15 mg BID (N=323)
Weight increased (Investigations) | 22 | 49 | 26 | 34
Dizziness (Nervous system disorders) | 17 | 56 | 47 | 36
Headache (Nervous system disorders) | 50 | 41 | 39 | 31
Somnolence (Nervous system disorders) | 9 | 40 | 29 | 39
Drug withdrawal syndrome (General disorders) | 10 | 12 | 15 | 21
Oedema peripheral (General disorders) | 4 | 18 | 11 | 15
Nausea (Gastrointestinal disorders) | 11 | 18 | 25 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 11 | 18 | 7
Urinary tract infection (Infections and infestations) | 14 | 10 | 20 | 16
Nasopharyngitis (Infections and infestations) | 13 | 19 | 13 | 14
Fatigue (General disorders) | 10 | 15 | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No